CLINICAL TRIAL: NCT05635305
Title: A Phase 1, Single-dose, Open-label, Randomized, 4-way Crossover Zoliflodacin Bioequivalence Study of the Reference Product (ZoliPa) With the Test Product (ZoliDr) in Healthy Adult Volunteers Under Fasted and Specific Fed Conditions Paired With an Investigation of the Effect of Cytochrome P450 3A4 Inhibition by Itraconazole on 3g Zoliflodacin (ZoliPa) Single-dose Pharmacokinetics
Brief Title: Zoliflodacin Bioequivalence and Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Antibiotics Research and Development Partnership (Other)
Collaborators: Parexel (Industry); KCAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STI_Zoli003
Record Dates: First submitted 2022-11-02; First posted 2022-12-02 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence; Drug Drug Interaction

STUDY DESIGN:
Intervention Model Description: BE study (cohort 1) will be managed in parallel with the DDI study (cohort 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BE study (Experimental): Cohort 1 (BE) is a four-period, four-sequence, four-treatment crossover BE and food effect study of zoliflodacin granules for oral suspension manufactured by Dr. Reddy's (test product, ZoliDr) and those manufactured by Patheon (reference product, ZoliPa) as a 3 g oral dose under fasting and a [specific] fed condition. This cohort will comprise of approximately 32 subjects (8 healthy subjects per treatment sequence) in 4 x 4 BE treatment arms in fasted and [specific] fed conditions. Healthy subjects will be randomized into 4 parallel treatment sequences to receive sequential Treatments A, B, C, and D in William's Square design pattern where:
  * Treatment A is ZoliPa fasted
  * Treatment B is ZoliDr fasted
  * Treatment C is ZoliPa [specific] fed condition
  * Treatment D is ZoliDr [specific] fed condition
  Based on William's Square design, below treatment sequences will be followed:
  A-B-C-D B-A-D-C C-D-A-B D-C-B-A
  Interventions: Drug: Zoliflodacin Patheon
- DDI study (Experimental): This is an open-label, 2-period, 2-treatment, fixed sequence crossover DDI study in healthy subjects. It will investigate PK of zoliflodacin (ZoliPa) in the absence and presence of itraconazole. Approximately 18 subjects will receive ZoliPa on Day 1 under fasting condition. After a washout of 72 hours after dosing of ZoliPa, on Day 4, subjects will receive a 400 mg loading dose of itraconazole followed by 200 mg of itraconazole once daily from Day 5-8. From Day 4 to Day 8, itraconazole will be administered immediately after a full meal. On Day 9, both itraconazole and zoliflodacin (ZoliPa) will be administered under fasting conditions at -1 hours and 0 hours, respectively. Itraconazole will then be administered with food at 24 hours (Day 10) and 48 hours (Day 11) after administration of zoliflodacin (ZoliPa).
  Interventions: Drug: Zoliflodacin Patheon

INTERVENTIONS:
Drug: Zoliflodacin Patheon — Zoliflodacin Patheon formulation to be compared with Zoliflodacin Dr Reddy's formulation during BE study (cohort 1).
  Itraconazole will be administered with Zoliflodacin Patheon formulation during DDI study (cohort 2)

SUMMARY:
this study will be a Phase 1, single-dose, two parallel cohorts, open-label, randomized study in healthy subjects with Cohort 1 as bioequivalence (BE) and food effect study and Cohort 2 as a drug-drug interaction (DDI) study.

DETAILED DESCRIPTION:
Cohort 1 (BE) is a four-period, four-sequence, four-treatment crossover BE and food effect study of zoliflodacin granules for oral suspension manufactured by Dr. Reddy's (test product, ZoliDr) and those manufactured by Patheon (reference product, ZoliPa) as a 3 g oral dose under fasting and a [specific] fed condition. This cohort will comprise of approximately 32 subjects (8 healthy subjects per treatment sequence) in 4 x 4 BE treatment arms in fasted and [specific] fed conditions. Healthy subjects will be randomized into 4 parallel treatment sequences to receive sequential Treatments A, B, C, and D in William's Square design pattern where:

* Treatment A is ZoliPa fasted
* Treatment B is ZoliDr fasted
* Treatment C is ZoliPa [specific] fed condition
* Treatment D is ZoliDr [specific] fed condition

Based on William's Square design, below treatment sequences will be followed:

A-B-C-D B-A-D-C C-D-A-B D-C-B-A

There will be 4 treatment periods, each with a single dose of the investigational medicinal products (IMP).

The washout period between each IMP administration will be at least 72 hours. Food regimen: Subjects, who are in a treatment period in which they are [specific] fed, will be dosed 30 minutes after the start of food intake. The subjects are expected to consume the entire meal within 30 minutes prior to dosing.

Cohort 2 (DDI): This is an open-label, 2-period, 2-treatment, fixed sequence crossover DDI study in healthy subjects. It will investigate PK of zoliflodacin (ZoliPa) in the absence and presence of itraconazole. Approximately 18 subjects will receive ZoliPa on Day 1 under fasting condition. After a washout of 72 hours after dosing of ZoliPa, on Day 4, subjects will receive a 400 mg loading dose of itraconazole followed by 200 mg of itraconazole once daily from Day 5-8. From Day 4 to Day 8, itraconazole will be administered immediately after a full meal. On Day 9, both itraconazole and zoliflodacin (ZoliPa) will be administered under fasting conditions at -1 hours and 0 hours, respectively. Itraconazole will then be administered with food at 24 hours (Day 10) and 48 hours (Day 11) after administration of zoliflodacin (ZoliPa).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, 18 to 55 years of age at the time of signing of informed consent.
2. Body mass index (BMI, Quetelet index, calculated as weight in kg/height in m2) between 18.0 and 30.0 kg/m2 (both inclusive) and weigh at least 50 kg and no more than 95 kg inclusive at Screening.
3. Healthy subjects, defined as individuals who are free from clinically significant illness or disease as determined by their medical/surgical history, normal vital signs, normal physical examination, normal standard 12-lead electrocardiogram (ECG), and laboratory investigations.
4. At the Screening visit, supine vital signs must be within the following ranges:

   * Systolic blood pressure (SBP) between 90 and 139 mmHg
   * Diastolic blood pressure (DBP) between 60 and 89 mmHg
   * Pulse between 50 and 90 beats per minute (bpm)
   * Tympanic temperature between 35.0 and 37.5°C Note: These will be measured after resting for 10 min.
5. Able to understand and communicate in German/or native language of the site with the Investigator and research staff and to comply with the requirements of the entire study. Provision of written informed consent to participate in the study.
6. Female subjects, if:

   o Not of childbearing potential, e.g., have a documentation of irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy and/or bilateral tubal ligation, at least 6 weeks before the Screening visit, amenorrhea for ≥ 12 months and follicle stimulating hormone (FSH) in the post menopausal range according to local laboratory ranges.

   o Of childbearing potential (for inclusion in Cohort 1, BE Study only), the following conditions are to be met: i. Negative pregnancy test: If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received zoliflodacin, the IMP, every attempt must be made to follow her to term and the newborn(s) up to 2 years of age.

   ii. Not lactating iii. The female subject must agree to use, with their partner, an approved method of highly effective contraception in combination with a barrier method from at least 1 month before the Screening visit until 1 month after last dosing of IMP. Female subjects must agree not to attempt to become pregnant, must not donate ova from the Screening visit until at least 1 month after last dosing of IMP.

   The following are considered to be highly effective methods of birth control:
   1. Hormonal contraception (i.e., combined oral contraceptives, injectable or implantable hormonal contraceptives
   2. Hormonal or non-hormonal intrauterine device/system with a proven failure rate <1%
   3. The subject's male partner has undergone confirmed effective surgical sterilization before the female subject entered the clinical study and he is the sole sexual partner of the female subject during the clinical study
   4. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation symptothermal, post ovulation methods], declaration of abstinence for the duration of the study and withdrawal are not acceptable methods of contraception).

   Barrier methods of contraception include:
   1. Condom (with or without spermicidal foam/gel/film/cream/ suppository but not use of fat/oil containing lubricants).
   2. Occlusive cap (diaphragm or cervical/vault caps) with spermicidal gel/film/cream/suppository.
   3. Other methods, if considered by the Investigator as reliable, will be accepted.
7. Male subjects who agree to use appropriate contraception methods to prevent pregnancy in their female partner(s) from the time of first dose until one month after last dose of IMP administration, i.e., condoms with or without spermicide. A male subject should be instructed that, unless his female partner(s) has had a tubal ligation, hysterectomy, or bilateral oophorectomy or is post-menopausal, his female partner(s) should use another form of contraception from the time of first dosing until one month after last dose of IMP administration - such other forms of contraception include an intrauterine device, condom, diaphragm with spermicide, oral contraceptive, injectable progesterone, or subdermal implant; male subjects who have been vasectomized at least 6 months before the first dose of IMP are exempt from the use of condom, and his female partner(s) do(es) not need any additional form of contraception.
8. Provision of written informed consent to participate in the study.
9. Subjects in the BE cohort must be willing to consume the meal prescribed with administration of the IMP in full and within the required time under fed conditions.

Exclusion Criteria:

1. For Cohort 2, DDI Study only: Female subjects of childbearing potential.
2. Subject has a positive RT PCR test for SARS-CoV-2 prior to randomization.
3. Subject has clinical signs and symptoms consistent with SARS-CoV-2 infection, e.g., fever, dry cough, dyspnea, sore throat, fatigue, or positive SARS-CoV-2 test result within 4 weeks prior to Screening.
4. Subject had severe course of COVID-19 (i.e., hospitalization, extracorporeal membrane oxygenation [ECMO], or mechanically ventilated) less than 3 months prior to Screening.
5. Subject received or is planning to receive a COVID-19 vaccine within 3 weeks prior to the first IMP administration until Post-study visit.
6. Recent (within previous 14 days) exposure to someone who has COVID-19 symptoms or positive test result.
7. Has a current occupation that involves routine exposure to potential COVID-19 patients or sources of SARS-CoV-2 (e.g., healthcare worker).
8. History of orthostatic hypotension (drop of >20 mmHg at systolic blood pressure, drop of > 10 at diastolic blood pressure, and/or heart rate increase of >30 bpm and >120 bpm after 3 minutes in standing position).
9. Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
10. History or presence of any clinically significant acute or chronic disease, including known or suspected human immunodeficiency virus (HIV), hepatitis A virus (HAV), HBV, or HCV infection (confirmed by positive laboratory test for anti-HAV IgM antibodies, hepatitis B surface antigen (HbsAg), or anti-HIV1/2 or anti-HCV antibodies).
11. Receipt of zoliflodacin, vaccines, biologics, or any other investigational product within 3 months prior to study start or during the study, or 5-times the half-life of the drug tested in the previous clinical study, whichever is longer (time calculated relative to the last dose in the previous clinical study). Influenza vaccination and SARS-CoV-2 vaccination prior to Screening will be allowed.
12. Presence of clinically significant abnormality following review of pre-study laboratory tests (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], or creatinine > upper limit of normal [ULN]), vital signs, full physical examination, and ECG.
13. History of serious allergy, allergic skin rash, history of drug allergy to itraconazole or other azole antifungals or allergy/sensitivity to any drug.
14. Excessive intake of caffeine (more than 8 cups daily of beverage containing caffeine).
15. Current alcohol use >21 units of alcohol per week for males and >14 units of alcohol per week for females (one unit = 8 g or about 10 mL of pure alcohol) and/or positive urine alcohol test at Screening.
16. Known or suspected drug abuse or positive laboratory test for urine drug screening (opiates, cocaine, amphetamine, cannabis, benzodiazepines).
17. Use of any medication, prescribed or over-the-counter (including antacid drug, except for acetaminophen [paracetamol up to 4 g/day]), or herbal remedies, during the 28 days before the first dose of IMP except if this will not affect the outcome of the study in the opinion of the Investigator.
18. Use of any enzyme-modifying drugs and/or other products, including strong or moderate inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong or moderate inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort and rifampicin) in the previous 30 days before first IMP administration until the last blood draw in the study.
19. Consumption of food or beverages containing grapefruit and/or pomelo within 14 days prior to first IMP administration until the last blood draw in the study.
20. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing until the last blood draw in the study.
21. Treatment within the previous 3 months before the first administration of IMP with any drug with a well defined potential for adversely affecting a major organ or system.
22. A major illness during the 3 months before commencement of the Screening period.
23. Presence of clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study.
24. Subjects who had abdominal surgery (e.g., gastric, small intestine or colon resection or bypass) or medical condition that might affect absorption of IMP taken orally.
25. History of gastrointestinal ulcer disease, inflammatory bowel disease, indigestion symptoms >3 times a week, or blood in stool in previous 6 months not related to anal trauma.
26. Who had febrile illness within 1 week before the start of the study.
27. Who has regular daily consumption of more than 1 L of xanthine containing beverages.
28. The subject has smoked, used tobacco products, e-cigarette or used nicotine replacement products within the 3 months before the first dosing or has a positive cotinine screen in urine.
29. Any clinically important abnormalities in heart rate, rhythm, conduction, or morphology of resting ECG that in the opinion of the Investigator are clinically significant or may interfere with the interpretation of QTc interval changes. QT interval corrected using QTcF >450 ms for male subjects and 460 ms for female subjects on Screening ECG. Clinically significant history or presence of myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval or conduction abnormalities.
30. History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
31. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
32. Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP or have donated plasma within 7 days of study dosing.
33. Clinically relevant abnormalities in the coagulation status or history of bleeding disorders.
34. Vulnerable subjects, e.g., persons in detention, protected adult under guardianship/trusteeship, soldier or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Cmax | through study completion, an average of 5 months
  Maximum observed plasma concentration
AUC(0-t) | through study completion, an average of 5 months
  Area under the plasma concentration versus time curve, from time zero to t, where t is the time of the last quantifiable concentration
AUC(0-∞) | through study completion, an average of 5 months
  Area under the plasma concentration versus time curve, with extrapolation to infinity
clinically significant changes from baseline for vital signs: HR | through study completion, an average of 5 months
  clinically significant changes from baseline for heart rate
clinically significant changes from baseline for vital signs: SBP | through study completion, an average of 5 months
  clinically significant changes from baseline for Systolic Blood Pressure
clinically significant changes from baseline for vital signs: DBP | through study completion, an average of 5 months
  clinically significant changes from baseline for Diastolic Blood Pressure
clinically significant changes from baseline for ECG: PR | through study completion, an average of 5 months
  clinically significant changes from baseline for PR
clinically significant changes from baseline for ECG: QRS | through study completion, an average of 5 months
  clinically significant changes from baseline for QRS
clinically significant changes from baseline for ECG: QTcF | through study completion, an average of 5 months
  clinically significant changes from baseline for QTcF
TEAE | through study completion, an average of 5 months
  drug-related treatment-emergent

SECONDARY OUTCOMES:
tmax | through study completion, an average of 5 months
  Time to maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Salman Nasr, MD, Principal Investigator — Parexel CPU Berlin, Germany
Locations (1):
- Parexel Early Phase Clinical Unit, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No